CLINICAL TRIAL: NCT04511364
Title: Long-term Follow-up in Osteoporotic Women Treated with Local Osteo-Enhancement in Europe
Brief Title: CONFIRM EXTENSION - Long-term Follow-up Study of Patients Treated with AGN1 LOEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AgNovos Healthcare, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AGN-CIP-300
Record Dates: First submitted 2020-08-04; First posted 2020-08-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Osteoporosis
Keywords: local osteo-enhancement procedure; hip fracture/prevention and control; calcium phosphate; calcium sulphate; LOEP; CONFIRM Extension
MeSH Terms: conditions — Osteoporosis; Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AGN1 treated patients (Experimental): Patients have been treated with the AGN1 LOEP kit in AgNovos study PST-EU-101.1. An X-ray and DXA scan are performed at 24 and 60 months post AGN1 LOEP treatment.
  Interventions: Other: Clinical imaging is performed during the 24 and 60 month follow-up visits

INTERVENTIONS:
Other: Clinical imaging is performed during the 24 and 60 month follow-up visits — X-ray and DXA scan

SUMMARY:
The study is designed as a multi-center study within Europe in up to 60 patients treated with the AGN1 LOEP Kit in CONFIRM. This will be a non-randomized and non-blinded study. The study will collect long-term follow-up data on the safety and clinical performance of AGN1 LOEP.

To qualify, subjects must have previously consented, enrolled, and been treated with the AGN1 LOEP kit in CONFIRM (AgNovos Study PST-EU-101.1).

Follow-up evaluations will be conducted at 24, 36, 48 and 60 months from the date the subject originally received the AGN1 LOEP treatment. Subjects will receive DXA and X-ray imaging at the 24- and 60-month follow-up visits. The 36- and 48-month follow-up evaluations will be conducted by phone. All timepoints will include general health and medical record review.

ELIGIBILITY:
Inclusion Criteria:

* Subject had previously enrolled in CONFIRM and received AGN1 LOEP treatment.
* Subject has willingness, ability, and commitment to participate in baseline and follow-up evaluations for the full length of the study.
* Subject is capable of giving written informed consent to participate in the study.

Exclusion Criteria:

* Subject was withdrawn from CONFIRM.
* Subject has severe comorbidity or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in DXA score at 24 months | 24 months
  Change in DXA score of treated hip from baseline pre-AGN1 LOEP to 24 months post-treatment.

SECONDARY OUTCOMES:
Change in DXA score at 60 months | 60 months
  Change in DXA score of treated hip from pre-AGN1 LOEP to 60 months post-treatment.
Hip fracture incidence | 60 months
  The incidence of hip fracture on the treated side during the follow-up period through 60 months post-AGN1 LOEP treatment.
Radiologic bone formation | 60 months
  Radiologic appearance of bone formation as assessed by X-ray at 24 and 60 months post-treatment.

OTHER OUTCOMES:
Safety evaluation | 60 months
  The incidence of all serious adverse events during follow-up determined to be at least possibly related to the procedure and/or device through 60 months post-AGN1 LOEP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jo De Schepper, MD, Principal Investigator — AZ Nikolaas
Locations (1):
- AZ Nikolaas, Sint-Niklaas, Sint-Niklaas, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pajor A, Grof J, Idei M, Menyhart J, Zsolnai B. Utero-inhibin: a new substance inhibiting uterine contraction, isolated from amniotic fluid. Acta Physiol Acad Sci Hung. 1982;59(4):325-8. PMID 7170985
- [Background] Harsoulis P, Ekonomou A, Leontsini M, Efthimiou E, Gerasimidis T, Vlotidis J, Sbarounis C. Fine needle aspiration biopsy cytology in the diagnosis of thyroid cancer. Acta Endocrinol Suppl (Copenh). 1984;265:50-1. doi: 10.1530/acta.0.107s0050. No abstract available. PMID 6593990